CLINICAL TRIAL: NCT07375706
Title: Clinical Performance of Posterior Resin Composite Restorations Placed by Undergraduate Students and Postgraduate Trainees: A Retrospective Study Using USPHS and FDI Criteria
Brief Title: Operator Experience and Restorative Clinical Performance of Posterior Composite Restorations
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Narmin Mammadli, DDS, Specialist in Pediatric Dentistry, Bezmialem Vakif University
Other Study IDs: 08.07.2024-E.157036
Record Dates: First submitted 2026-01-13; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Dental Restoration Failure
Keywords: Pediatric Dentistry; USPHS Criteria; FDI Criteria; Operator Experience; Dental Restoration Longevity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Undergraduate Operators: Posterior resin composite restorations placed by undergraduate dental students as part of routine clinical training in the Department of Pediatric Dentistry. All restorations were performed under faculty supervision and evaluated retrospectively using standardized clinical assessment criteria.
- Postgraduate Operators: Posterior resin composite restorations placed by postgraduate specialty trainees in pediatric dentistry during routine clinical care. Restorations were retrospectively evaluated using the same clinical assessment protocols as the undergraduate group.

SUMMARY:
This retrospective observational study aimed to evaluate the long-term clinical performance of posterior resin composite restorations placed by undergraduate dental students and postgraduate specialty trainees in pediatric patients. Dental records of children aged 6 to 13 years who received posterior composite restorations at a university-based pediatric dentistry clinic were reviewed.

A total of 200 restorations placed on primary and permanent molars were clinically evaluated during routine follow-up visits using standardized assessment systems. The modified United States Public Health Service (USPHS) criteria and the FDI World Dental Federation criteria were used to assess esthetic, functional, and biological outcomes. Evaluations were performed by a blinded examiner, and radiographic assessments were conducted when clinically indicated.

Clinical outcomes were compared between operator groups according to training level, follow-up duration, restoration type, tooth type, and endodontic treatment history. The findings of this study aim to provide insight into the impact of operator experience on the clinical success and longevity of posterior resin composite restorations in pediatric dentistry and to support evidence-based improvements in undergraduate and postgraduate dental education.

DETAILED DESCRIPTION:
This retrospective observational study was conducted at the Department of Pediatric Dentistry of a university-based dental faculty to compare the clinical performance of posterior resin composite restorations placed by undergraduate dental students and postgraduate specialty trainees.

Dental records of pediatric patients aged 6 to 13 years who received posterior resin composite restorations on primary or permanent first and second molars were retrospectively reviewed. A total of 200 restorations were included in the study, of which 100 were placed by undergraduate students and 100 by postgraduate trainees. All restorations were placed using the same microhybrid resin composite material as part of routine clinical care.

Restorations were excluded if they were placed by operators outside the defined study groups, if materials other than resin composite were used, if follow-up duration was less than three months, or if the restorations were placed on teeth other than posterior molars. Clinical evaluations were performed during routine follow-up or concurrent dental treatment visits.

All restorations were assessed by a blinded examiner using two standardized evaluation systems: the modified United States Public Health Service (USPHS-Ryge) criteria and the FDI World Dental Federation (FDI-Hickel) criteria. Esthetic, functional, and biological parameters were evaluated clinically, and radiographic assessments were performed when clinically indicated. Under the USPHS criteria, restorations were categorized as acceptable or unacceptable. According to the FDI criteria, scores of 1-2 were considered successful, score 3 clinically acceptable, and scores of 4-5 unsuccessful.

Recorded variables included operator group, restoration type (one-, two-, or three-surface), follow-up duration, tooth type (primary or permanent), patient age, and endodontic treatment history. Clinical outcomes were compared between operator groups and across follow-up intervals to evaluate the influence of operator experience and time on restoration performance.

Statistical analyses were performed using appropriate non-parametric tests due to non-normal data distribution. Descriptive statistics were used to summarize the data, and group comparisons were conducted with a significance level set at p < 0.05.

The results of this study aim to clarify the role of operator experience in the long-term success of posterior resin composite restorations in pediatric patients and to contribute to evidence-based improvements in undergraduate and postgraduate dental training programs.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 13 years at the time of treatment
* Patients who received posterior resin composite restorations on primary or permanent first or second molars
* Restorations placed by undergraduate dental students or postgraduate specialty trainees in the Department of Pediatric Dentistry
* Restorations with a minimum follow-up period of 3 months
* Availability of complete clinical records allowing retrospective evaluation

Exclusion Criteria:

* Restorations placed by clinicians outside the undergraduate or postgraduate trainee groups
* Restorations performed using materials other than resin composite
* Restorations placed on teeth other than posterior molars
* Restorations with a follow-up duration shorter than 3 months
* Incomplete or missing clinical records preventing standardized evaluation

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population consisted of children aged 6 to 13 years who received posterior resin composite restorations on primary or permanent molar teeth at a university-based pediatric dentistry clinic. All included restorations were placed by undergraduate dental students or postgraduate specialty trainees as part of routine clinical care. Patients were identified retrospectively through institutional dental records, and only cases with sufficient clinical documentation and a minimum follow-up period of three months were included for evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2025-01-23 (Actual); Study Completion 2025-02-17 (Actual)

PRIMARY OUTCOMES:
Clinical Performance of Posterior Resin Composite Restorations Assessed by Modified USPHS-Ryge Criteria | Up to 24 months
  The clinical performance of posterior resin composite restorations was evaluated using the modified United States Public Health Service (USPHS-Ryge) criteria. Based on esthetic, functional, and biological parameters, restorations were categorized into two groups according to clinical acceptability: acceptable (+) and unacceptable (-).
Clinical Performance of Posterior Resin Composite Restorations Assessed by FDI World Dental Federation Criteria | Up to 24 months
  The clinical performance of posterior resin composite restorations was evaluated using the FDI World Dental Federation (Hickel) criteria, based on esthetic, functional, and biological parameters. Restorations were scored on a 5-point ordinal scale ranging from 1 to 5, where scores of 1 and 2 were considered successful, score 3 clinically acceptable, and scores of 4 and 5 unsuccessful. Higher scores indicate worse clinical performance.

SECONDARY OUTCOMES:
Comparison of Clinical Performance Between Undergraduate and Postgraduate Operators Using USPHS Criteria | Up to 24 month
  Clinical performance outcomes assessed by the modified USPHS-Ryge criteria were compared between undergraduate dental students and postgraduate specialty trainees across follow-up periods.
Comparison of Clinical Performance Between Undergraduate and Postgraduate Operators Using FDI Criteria | Up to 24 month
  Clinical performance outcomes assessed by the FDI World Dental Federation criteria were compared between undergraduate dental students and postgraduate specialty trainees across follow-up periods.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakıf University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because this study is a retrospective observational study involving pediatric patients, and data use is restricted by ethical approval and institutional policies. In addition, informed consent for data sharing beyond the scope of the original study was not obtained, and all analyses were conducted using anonymized clinical records.